CLINICAL TRIAL: NCT02412865
Title: Developing and Scaling a Text Messaging Tool to Help Pregnant Smokers
Brief Title: Quit4Baby Evaluation
Acronym: Quit4Baby
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Responsible Party: Principal Investigator, Lorien Abroms, Associate Professor, George Washington University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R44 DA035017-0 2; R44DA035017 (NIH)
Record Dates: First submitted 2015-03-31; First posted 2015-04-09 (Estimated); Last update posted 2016-02-26 (Estimated); Status verified 2016-02

CONDITIONS: Smoking Cessation; Pregnancy
Keywords: mhealth
MeSH Terms: conditions — Smoking Cessation

ARMS (2):
- Intervention (Experimental): quit4baby + text4baby
  Interventions: Behavioral: Quit4Baby; Behavioral: Text4Baby
- Control (Other): text4baby
  Interventions: Behavioral: Text4Baby

INTERVENTIONS:
Behavioral: Quit4Baby
  Arms: Intervention
Behavioral: Text4Baby

SUMMARY:
The goal of this project is to evaluate the effectiveness (Phase II) of a text-based program to be called Quit4Baby to support smoking cessation efforts of pregnant women who smoke.

In Phase II, Dr. Abroms will conduct a randomized clinical trial among 500 pregnant smokers who have been recruited from users of text4baby - the first large scale mobile health application in the United States. Developed and operated by Voxiva and Healthy Mothers, Healthy Babies (HMHB)-collaborators in this program -text4baby is a free national service that has enrolled more than 800,000 pregnant women and mothers of infants 0-1 nationwide and delivered more than 150 million health messages to them including messages encouraging them not to smoke during pregnancy and referring them to quit lines.

Hypothesis 1: Pregnant smokers who receive quit4Baby + text4Baby will demonstrate higher levels of knowledge about the dangers of second hand smoke and the benefits of smoking cessation for mothers and their infants than text4baby only users.

Hypothesis 2: Pregnant smokers who receive quit4baby + text4baby will report significantly higher rates of calling a quit line, discussions with their health provider and/or use of cessation counseling than those who receive Text4baby alone.

Hypothesis 3: Pregnant smokers who receive quit4baby + text4baby will have significantly more favorable quitting outcomes compared with text4baby alone.

ELIGIBILITY:
Inclusion Criteria:

1. Subscribe to the text4baby test messaging program
2. Pregnant
3. Smoke or recently quit (within last 2 weeks)- Smoking will be defined as self-report of smoking at least one cigarette in the past 7 days. Given that these individuals are recruited from text4baby users, we are confident that they will have cell phones and text messaging capacity.
4. Speak English
5. Willing to enroll in our study
6. 14 years old or older

Exclusion Criteria:

1. No longer subscribe to text4baby
2. Not pregnant
3. Not current smoker (within past 2 weeks)
4. Non-English speakers
5. Not willing to receive Quit4Baby messages or enroll in study
6. Younger than 14 years of age

Ages: 14 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 505 (Actual)
Dates: Start 2015-04; Primary Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Biometrically confirmed abstinence | 3-6 months
  With saliva cotinine
Quitline call rates | 1-6 months
Knowledge as measured by survey items | 1-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- The George Washington University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Abroms LC, Johnson PR, Heminger CL, Van Alstyne JM, Leavitt LE, Schindler-Ruwisch JM, Bushar JA. Quit4baby: results from a pilot test of a mobile smoking cessation program for pregnant women. JMIR Mhealth Uhealth. 2015 Jan 23;3(1):e10. doi: 10.2196/mhealth.3846. PMID 25650765
- [Derived] Palmer MJ, Henschke N, Bergman H, Villanueva G, Maayan N, Tamrat T, Mehl GL, Glenton C, Lewin S, Fonhus MS, Free C. Targeted client communication via mobile devices for improving maternal, neonatal, and child health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013679. doi: 10.1002/14651858.CD013679. PMID 32813276